CLINICAL TRIAL: NCT04951258
Title: Effect of Multicomponent Exercise on Cognitive Function and Activities of Daily Living in People With Dementia
Brief Title: Multicomponent Exercise in People With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM110062F
Record Dates: First submitted 2021-06-18; First posted 2021-07-06 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent exercise group (Experimental)
  Interventions: Other: Multicomponent exercise
- Video home exercise group (Active Comparator)
  Interventions: Other: Video home exercise group

INTERVENTIONS:
Other: Multicomponent exercise — The intervention is a 60-minute session, 3 times/week, totaling 9 weeks. Multicomponent exercise included strengthening, balance training, aerobic dance, and stretching
  Arms: Multicomponent exercise group
Other: Video home exercise group — The intervention is a 60-minute session, 3 times/week, totaling 9 weeks. Video home exercise included four limbs mobility exercise, stretching, strengthening, and aerobic exercise
  Arms: Video home exercise group

SUMMARY:
People with dementia shows a decline in cognition, such as memory, executive function (EF), language, attention, and spatial orientation that is significant enough to interfere with the independence and daily functioning. Previous studies reported that multicomponent exercise improved EF in people with mild cognitive impairment and independence of ADL in those with Alzheimer's disease. However, few studies investigated whether multicomponent exercise improved EF, memory, and ADL in people with dementia. Therefore, the purposes of this study are to examine 1) the effect of multicomponent exercise on EF, memory, and ADL in people with mild to moderate dementia; 2) the correlation between change in EF and ADL; 3) the correlation between change in memory and ADL.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60-80 y/o
* Mini-Mental State Examination: 10-26
* Clinical Dementia Rating: 1-2
* Walk at least 6 meters independently (with or without walking aids)

Exclusion Criteria:

* Any other diagnosis of neurological diseases or musculoskeletal problems (Except dementia)
* Physical or psychological comorbidities that affect performance during assessment or intervention
* Already participating in other physical training in the last 1 month

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | Change from baseline at 9 week
  It is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Higher scores mean a better outcome.
Chinese version of Verbal learning test | Change from baseline at 9 week
  It is a 9-point measurement to evaluate memory. Higher scores mean a better outcome.
Chinese version of Stroop color and word test | Change from baseline at 9 week
  It is a measurement to evaluate inhibition control.
Digit span test | Change from baseline at 9 week
  It is a measurement to evaluate working memory.
Trail making test - Chinese version | Change from baseline at 9 week
  It is a measurement to evaluate cognitive flexibility.

SECONDARY OUTCOMES:
Barthel index | Change from baseline at 9 week
  It is a 100-point ordinal scale used to measure performance in activities of daily living. Higher scores mean a better outcome.
Instrumental activities of daily living (IADL) scale | Change from baseline at 9 week
  It is a 24-point ordinal scale used to measure performance in instrumental activities of daily living. Higher scores mean a better outcome.
Chinese version of Quality of Life in Alzheimer Disease Scale | Change from baseline at 9 week
  It is a measurement to evaluate quality of life. The scale scores range from 13 to 52, with higher scores indicating greater quality of life.
Time up and go test | Change from baseline at 9 week
  It is a test to evaluate functional mobility.
30-second chair stand test | Change from baseline at 9 week
  It is a test to evaluate muscle strength.
6-minute walk test | Change from baseline at 9 week
  It is a test to evaluate endurance.
Berg Balance Scale | Change from baseline at 9 week
  It is a tool to evaluate balance. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.

IPD SHARING:
Plan to Share IPD: Undecided